CLINICAL TRIAL: NCT04620187
Title: A Phase II Study of Adjuvant Ado-trastuzumab Emtansine (T-DM1) in HER2-positive Salivary Gland Carcinomas
Brief Title: Post-op T-DM1 in HER-2+ Salivary Gland Carcinomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-432
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Salivary Gland Cancer; HER2 Gene Mutation
Keywords: Salivary Gland Cancer; HER2 Gene Mutation
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Maytansine; Ado-Trastuzumab Emtansine; Radiation; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard of Care + T-DM1 in HER2-Positive Salivary Gland Cancer (Experimental): Participants will undergo standard of care surgery followed by standard of care radiation and chemotherapy with the addition of T-DM1.
  Study cycles are 21 days (3 weeks):
  * Participants will be given the study treatment T-DM1 at a predetermined dose (3.6 mg/kg) intravenously once (1x) every 3 weeks for up to 52 weeks (or about 1 year).
  * Participants will be given standard of care radiation and chemotherapy
    * Radiation will be given on Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 2 Day 15, and Cycle 3 Day 1
    * Chemotherapy (cisplatin 40 mg/m2 intravenously or carboplatin AUC 2 intravenously) will be given on Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 2 Day 15, and Cycle 3 Day 1
  Participants will be followed for 3 years.
  Interventions: Drug: Ado-trastuzumab (T) emtansine (T-DM1); Radiation: Standard of Care Radiotherapy; Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Drug: Ado-trastuzumab (T) emtansine (T-DM1) — Intravenous infusion ever 21 days (3weeks) for 1 year (52 weeks)
  Other Names: Kadcyla
Radiation: Standard of Care Radiotherapy — Radiotherapy to shrink or kill tumors
  Other Names: Radiation
Drug: Standard of Care Chemotherapy — Intravenous injection
  Other Names: Cisplatin; carboplatin

SUMMARY:
This research is being done to see how safe and effective the use of the study drug Ado-trastuzumab (T) emtansine (DM1), T-DM1, and standard of care chemoradiation are when used together in treating HER2-positive salivary gland cancer. It will also examine the effectiveness of study drug Ado-trastuzumab (T) emtansine (DM1) on cancer recurrence.

DETAILED DESCRIPTION:
This is a phase II, open-label, non-randomized, multi-institutional study investigating postoperative or adjuvant human epidermal growth factor receptor (HER2)-directed therapy with adjuvant ado-trastuzumab emtansine (T-DM1) in HER2-positive salivary gland carcinomas (SGC).

This research study is:

* Studying the use of T-DM1 in combination with radiation and chemotherapy; and the use of maintenance T-DM1 alone for up to a year after surgery
* Evaluating the effectiveness, safety, and toxicity of T-DM1

T-DM1 is a specialized antibody targeting HER-2 (a protein that is expressed in some breast and salivary gland cancers). The drug is a HER-2 antibody that is bound to a chemotherapy agent (DM1) and delivered intravenously. T-DM1 then binds cancer cells that express HER-2 and is taken up into the cell to allow DM1 to kill cancer cells in a more targeted way. This allows the use of a targeted treatment along with chemoradiation to treat HER-2 expressing salivary cancers.

The U.S. Food and Drug Administration (FDA) has not approved T-DM1 for HER2-positive salivary gland cancer but it has been approved for other uses (for breast cancers that express HER2 protein).

The research study procedures include: screening for eligibility and study treatment including evaluations and follow up visits.

This research study involves radiation, chemotherapy, and targeted therapy given after surgery for up to 1-year, and participants will be followed for 3 years.

It is expected that about 55 people will take part in this research study.

Genentech is supporting this research study by providing the research study drug, T-DM1.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically or cytologically confirmed, resectable stage II (with positive margins), III, IVA, or IVB locoregionally advanced salivary gland carcinoma (including any histologic subtype), as defined by 2017 American Joint Committee on Cancer (AJCC), 8th edition.
* Willing to provide tissue from a diagnostic biopsy or at the time of cancer resection, and blood samples before, during, and after treatment.
* HER2 positive disease as defined by any of the following:

  * Tumor HER2 expression staining intensity of 2 or 3+ by IHC (from either a preoperative biopsy or resection specimen at the time of oncologic surgery)
  * HER2 amplification as determined by FISH (HER2/CEP 17 ratio greater than or equal to 2.0 or HER2 mean copy number greater than or equal to 4.0)
  * HER2 or ERBB2 mutated on tumor genomic sequencing assay (see Section 9.1 for permitted HER2 mutations)
* Age 18 years or older
* ECOG performance status ≤ 1 (Karnofsky ≥ 60%, see Appendix A)
* Participant must have normal organ and marrow function as defined below within 14 days prior to study registration:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,000/mcL
  * hemoglobin ≥ 9.0 g/dL
  * platelets ≥ 100,000/mcL
  * total bilirubin ≤ 2.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5× institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Serum calcium (corrected for albumin value), magnesium, and potassium levels within normal limits per institutional standards.
* Assessment of cardiac function either by an echocardiogram or a multi-gated acquisition (MUGA) scan prior to the therapy initiation, with a baseline left systolic ventricular ejection fraction (LVEF) ≥ 50% within 1 month prior to study registration.
* Ability to understand and the willingness to sign a written informed consent document.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of T-DM1. "Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 6 months after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception. See Appendix B for further guidance on contraception.

Exclusion Criteria:

* Patient with AJCC 2017 8th edition stage I or stage IVC (metastatic) disease, or unresectable disease.
* Subject who has had prior radiation and/or chemotherapy for head and neck cancer.
* Any history of prior HER2 directed therapy.
* Active or uncontrolled infection.
* Pregnant or lactating women.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has a known additional malignancy that is progressing or requires active treatment.

Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and low risk prostate adenocarcinoma being managed with active surveillance. A history of another separate malignancy in remission without evidence of active disease in the last 2 years is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
2 Year Disease-free survival (DFS) Rate | Time from the date of study registration to first invasive local, regional, distant recurrence, or death due to any cause assessed up to 36 months
  Kaplan-Meier method will be used to estimate 2 Year Disease-free survival (DFS) Rate

SECONDARY OUTCOMES:
Adverse Events | Time from study registration to death due to any cause, or censored at date last known alive assessed up to 36 months
  Evaluate adverse events for patient receiving T-DM1, defined as adverse events of all grades utilizing CTCAE v5
Overall survival (OS) Rate | Time from study registration to death due to any cause, or censored at date last known alive assessed up to 36 months
  Overall Survival (OS) estimated using a Kaplan-Meier or competing risk methodology (whichever is appropriate).
Distant metastatic-free survival (DMFS) Rate | Time from study registration to the earlier of the first occurrence of distant or metastatic disease, or death due to any cause assessed up to 36 months
  Distant metastatic-free survival (DMFS) Rate estimated using a Kaplan-Meier or competing risk methodology (whichever is appropriate).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - University of Chicago, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu